CLINICAL TRIAL: NCT05186350
Title: Comparison of SpyGlass Guided Lithotripsy Versus Extracorporeal Shockwaves Lithotripsy for Large Common Bile Duct Stones
Brief Title: SpyGlass Versus ESWL for Large Common Bile Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Professor, First People's Hospital of Hangzhou
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-01-06
Record Dates: First submitted 2022-01-06; First posted 2022-01-11 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Choledocholithiasis; Common Bile Duct Calculi
Keywords: Choledocholithiasis; SpyGlass; ESWL;ERCP
MeSH Terms: conditions — Choledocholithiasis; Gallstones

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SpyGlass group (Active Comparator): ERCP plus SpyGlass group
  Interventions: Procedure: ERCP+ SpyGlass
- ESWL group (Active Comparator): ERCP plus ESWL
  Interventions: Procedure: ESWL+ ERCP

INTERVENTIONS:
Procedure: ERCP+ SpyGlass — SpyGlass direct Vision guided laser lithotripsy
  Arms: SpyGlass group
Procedure: ESWL+ ERCP — ESWL + Stone removal through ERCP
  Arms: ESWL group

SUMMARY:
Overall stone clearance with endoscopic retrograde cholangiopancreatography (ERCP) for choledocholithiasis is a big problem, especially for stones with a diameter greater than 3cm. After ERCP failure, surgery was the option but patients not suitable for surgery were treated through stenting but had to undergo multiple ERCPs and show a success rate of only 44-96%. Recently, choledochoscopic laser, electrohydraulic lithotripsy, SpyGlass, or extracorporeal shock wave lithotripsy (ESWL) have been applied for the treatment of huge bile duct stones. The present study aims to compare the efficacy and safety outcomes of SpyGlass direct vision lithotripsy and ESWL procedures for the removal of large bile duct stones.

DETAILED DESCRIPTION:
ESWL was first used for the removal of renal calculi and ureteral calculi however, now a day is being used for biliary calculi. It has the advantages of simple operation, low cost, and higher safety. Recent studies show that the procedure time for ESWL is also shorter and the utilization rate of mechanical lithotripsy was effectively reduced with fewer complications. But It is difficult for ESWL to break the stones larger than 3cm into small pieces. So SpyGlass-guided laser lithotripsy is used. Spyglass has been used in clinics for more than ten years. Recently, a study reported difficult bile duct stones that were treated with SpyGlass-guided laser lithotripsy that shows promising results. Compared with laser lithotripsy under X-ray monitoring, there is no significant difference in stone removal rate and complication rate between the two methods. However, the effect of lithotripsy under Spyglass direct vision is better, which can break large stones into smaller pieces, thus making it easier to take stones. The investigators conducted the current study to compare the therapeutic outcome and complications between SpyGlass direct vision lithotripsy and ESWL procedures for the removal of large bile duct stones

ELIGIBILITY:
Inclusion Criteria:

* large bile duct stones (≥10 mm)

Exclusion Criteria:

* pregnancy
* refusal of written informed consent
* Patients with benign or malignant biliary stricture
* Contraindications to ERCP exist
* Complicated with acute pancreatitis or acute cholangitis
* Coagulation dysfunction#thrombocytopenia
* Patients after gastrointestinal reconstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Clearance rate(percentage) | 1 month
  Stone clearance ratio
Number of sessions | 1 month
  Number of ERCP procedures

SECONDARY OUTCOMES:
Complications | 1 month
  Side effect of the procedures
Procedure Time | Intraoperative
  Time spent for each surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Yang, Doctor, Principal Investigator — Affilated Hangzhou First People Hospital
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tao T, Zhang M, Zhang QJ, Li L, Li T, Zhu X, Li MD, Li GH, Sun SX. Outcome of a session of extracorporeal shock wave lithotripsy before endoscopic retrograde cholangiopancreatography for problematic and large common bile duct stones. World J Gastroenterol. 2017 Jul 21;23(27):4950-4957. doi: 10.3748/wjg.v23.i27.4950. PMID 28785149
- [Background] [French comment on article Cholangioscopy-guided lithotripsy for difficult bile duct stone clearance in a single session of ERCP: results from a large multinational registry demonstrate high success rates]. Endoscopy. 2019 Oct;51(10):1006-1007. doi: 10.1055/a-1000-5911. Epub 2019 Sep 26. No abstract available. French. PMID 31557778
- [Background] Manes G, Paspatis G, Aabakken L, Anderloni A, Arvanitakis M, Ah-Soune P, Barthet M, Domagk D, Dumonceau JM, Gigot JF, Hritz I, Karamanolis G, Laghi A, Mariani A, Paraskeva K, Pohl J, Ponchon T, Swahn F, Ter Steege RWF, Tringali A, Vezakis A, Williams EJ, van Hooft JE. Endoscopic management of common bile duct stones: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2019 May;51(5):472-491. doi: 10.1055/a-0862-0346. Epub 2019 Apr 3. PMID 30943551
- [Derived] Khizar H, Gu W, Zhou H, Yang J, Jin H, He X, Zhang X, Yang J. A comparative study of extracorporeal shock wave lithotripsy and cholangioscopy-guided lithotripsy in the management of complex biliary stones: A randomized trial. J Trauma Acute Care Surg. 2025 Oct 1;99(4):628-634. doi: 10.1097/TA.0000000000004693. Epub 2025 Aug 13. PMID 40811584